CLINICAL TRIAL: NCT04785651
Title: Evaluation of the Use of Tranexamic Acid in Tibial Osteotomies: a Randomised Controlled Clinical Trial.
Brief Title: Evaluation of the Use of Tranexamic Acid in Tibial Osteotomies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patient enrollment was proceeding slower than planned
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TXA-HTO
Record Dates: First submitted 2021-02-16; First posted 2021-03-08 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Monocompartimental Tibiofemoral Osteoarthritis; Osteoarthritis
Keywords: tibial osteotomy; tranexamic acid
MeSH Terms: conditions — Osteoarthritis | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic arm (Experimental): Patients in this arm will undergo to a tibial osteotomy in combination with the anti-fibrinolytic agent Tranexamic acid.
  Interventions: Drug: Tibial osteotomy with Tranexamic acid
- control arm (Other): Patients in this arm will undergo to a tibial osteotomy without the use of Tranexamic acid
  Interventions: Procedure: Tibial osteotomy without Tranexamic acid

INTERVENTIONS:
Drug: Tibial osteotomy with Tranexamic acid — Patients who will be in the treatment arm after randomisation will receive 100ml saline with a dosage of 20 mg/kg tranexamic acid intravenously at induction. An additional administration of tranexamic acid (10 mg/kg in 100ml intravenous saline) will be given as a booster at the end of the surgical procedure.
  All the patients will undergo to the same tibial osteotomy procedure.
  Arms: Tranexamic arm
Procedure: Tibial osteotomy without Tranexamic acid — Patients in this arm will undergo to the tibial osteotomy procedure as by clinical practice
  Arms: control arm

SUMMARY:
A randomised controlled double-blind clinical trial focused on the evaluation of the effectiveness of the tranexamic acid on bleeding, pain and wound complications reduction in tibial osteotomies.

All the 84 included patients will be randomized in one of the two arms, will undergo to a tibial osteotomy and then will prospectively evaluate at different follow ups until 60 days post-surgery

DETAILED DESCRIPTION:
Tibial osteotomies represents a well-established treatment option for the medial femorotibial knee arthrosis.

Osteotomy can be performed in minus or in plus, at the latter case with or without interposition of tissue (autologous bone, heterologous bone or bone substitute).

Even though excessive bleeding is not a frequent complication, the blood loss and formation of subcutaneous haematoma can determinate more post-interventional pain, wound suffering and the risk of infections.

Tranexamic acid is an antifibrinolytic agent and its use in proximal tibia osteotomies has been retrospectively evaluated in a number of papers, all of which agree on its safety and efficacy in terms of reducing peri-operative bleeding. However, to date there have been no randomised clinical trials demonstrating its superiority in terms of reducing bleeding, subcutaneous haematoma and wound complications in proximal tibia osteotomies.

This is a randomised controlled double-blind clinical trial focused on the evaluation of the effectiveness of the tranexamic acid on bleeding , pain and wound complications reduction in tibial osteotomies

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged between 18 and 70 years;
2. Single-part tibiofemoral osteoarthritis (K-L 1-3), axial deviation > 5°;
3. Surgical indication for corrective osteotomy;
4. Isolated osteotomy surgical procedure.

Exclusion Criteria:

1. Contraindication criteria for the administration of tranexamic acid, as assessed by the Anaesthesia and Resuscitation specialist during the pre-operative visit. The following will be considered absolute contraindications: epilepsy, thrombophilia and known allergy to the active substance, severe renal insufficiency and acute venous or arterial thrombosis, while the following will be considered relative contraindications: coronary stents in patients who have discontinued treatment with antiplatelet agents and previous deep vein thrombosis;
2. Known pro-thrombotic conditions (coagulation factor mutations, pregnancy status, previous pulmonary thromboembolism);
3. BMI > 40;
4. Incapacitated patients;
5. Patients abusing alcoholic beverages, drugs or medication.
6. Patients who are pregnant or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Perioperative blood loss (haemoglobin balance): | Basal vs the first post operative day
  The perioperative blood loss will be estimated by assessing the haemoglobin balance on the first postoperative day

SECONDARY OUTCOMES:
Postoperative transfusion rate | Perioperative time and postoperative time ( up to 60 days)
  the percentage of transfusions carried out in the two treatment groups will be determined;
Postoperative blood loss | Postoperatively (up to 2 days)
  The perioperative blood loss will be estimated by assessing the blood loss after surgery (through the volume of blood collected by drainage);
Blood loss after discharge | at 5 and 15 days post hospital discharge
  Post-discharge blood loss will be estimated by assessing haemoglobin balance at 5 and 15 days post-surgery;
International Knee Documentation Committee objective | Baseline, 30 and 60 days post treatment
  The objective rating scale has seven parameters related to knee function. The presence of effusions and degree of knee movement are assessed, the worst value of one of these parameters determines the final IKDC grade. There are four grades (A, B, C, D) that identify a knee assessed as normal, near normal, abnormal and severely abnormal, respectively.
Visual Analogue Scale - Pain | baseline, 1 day post-treatment, 2 days post-treatment, 1 month, 2 months);
  visual analogue scale consisting of a straight line segment (10 cm long), the ends of which correspond to 'no pain' and 'strongest pain imaginable'.
Soft tissue status | perioperatively, 30 and 60 days
  The condition of the soft tissues (swelling, surgical haematoma, wound distress) will be documented and analysed between the two groups by means of photographic documentation and through the Hollander Wound Evaluation Scales

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hunt BJ. The current place of tranexamic acid in the management of bleeding. Anaesthesia. 2015 Jan;70 Suppl 1:50-3, e18. doi: 10.1111/anae.12910. PMID 25440395
- [Background] Charoencholvanich K, Siriwattanasakul P. Tranexamic acid reduces blood loss and blood transfusion after TKA: a prospective randomized controlled trial. Clin Orthop Relat Res. 2011 Oct;469(10):2874-80. doi: 10.1007/s11999-011-1874-2. Epub 2011 Apr 22. PMID 21512813
- [Background] Palanisamy JV, Das S, Moon KH, Kim DH, Kim TK. Intravenous Tranexamic Acid Reduces Postoperative Blood Loss After High Tibial Osteotomy. Clin Orthop Relat Res. 2018 Nov;476(11):2148-2154. doi: 10.1097/CORR.0000000000000378. PMID 29939895